CLINICAL TRIAL: NCT02524951
Title: A Phase I Study of the Safety and Tolerability of Single Agent MSI-1436C in Metastatic Breast Cancer Patients
Brief Title: Safety and Tolerability of MSI-1436C in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of interest by sponsor
Sponsor: Northwell Health (Other)
Collaborators: DepYmed Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Budman, Director Translational Research, Cancer Institute, Northwell Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-0039
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 3-N-1(spermine)-7, 24-dihydroxy-5-cholestane 24-sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- MSI-1436C (Trodusquemine) 20 mg/m2 IV (Experimental): Open label, interventional, dose escalation of MSI-1436 (Trodusquemine), single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will receive MSI-1436 at a dose of 20 mg/m2. Drug infusions will last approximately 2 hours.
  Interventions: Drug: MSI-1436C
- MSI-1436C (Trodusquemine) 26 mg/m2 IV (Experimental): Open label, interventional, dose escalation of MSI-1436 (Trodusquemine), single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will receive MSI-1436 at a dose of 26 mg/m2. Drug infusions will last approximately 2 hours.
  Interventions: Drug: MSI-1436C
- MSI-1436C (Trodusquemine) 34 mg/m2 IV (Experimental): Open label, interventional, dose escalation of MSI-1436 (Trodusquemine), single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will receive MSI-1436 at a dose of 34 mg/m2 . Drug infusions will last approximately 2 hours.
  Interventions: Drug: MSI-1436C
- MSI-1436C (Trodusquemine) 44 mg/m2 IV (Experimental): Open label, interventional, dose escalation of MSI-1436 (Trodusquemine), single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will receive MSI-1436 at a dose of 44 mg/m2 . Drug infusions will last approximately 2 hours.
  Interventions: Drug: MSI-1436C
- MSI-1436C (Trodusquemine) 57 mg/m2 IV (Experimental): Open label, interventional, dose escalation of MSI-1436 (Trodusquemine), single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will receive MSI-1436 at a dose of 57 mg/m2. Drug infusions will last approximately 2 hours.
  Interventions: Drug: MSI-1436C
- MSI-1436C (Trodusquemine) 74 mg/m2 IV (Experimental): Open label, interventional, dose escalation of MSI-1436 (Trodusquemine), single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will receive MSI-1436 at a dose of 74 mg/m2 . Drug infusions will last approximately 2 hours.
  Interventions: Drug: MSI-1436C
- MSI-1436C (Trodusquemine) 96 mg/m2 IV (Experimental): Open label, interventional, dose escalation of MSI-1436 (Trodusquemine), single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will receive MSI-1436 at a dose of 96 mg/m2 . Drug infusions will last approximately 2 hours.
  Interventions: Drug: MSI-1436C

INTERVENTIONS:
Drug: MSI-1436C — Dose escalation, single intravenous infusion twice a week for 3 weeks on a 4-week cycle.
  Other Names: Trodusquemine

SUMMARY:
This is a Phase I, open-label, dose escalation study. MSI-1436 will be administered as a single intravenous infusion twice a week for 3 weeks on a 4-week cycle.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose escalation study. MSI-1436 will be administered as a single intravenous infusion twice a week for 3 weeks on a 4-week cycle. Subjects will be enrolled according to a standard Phase I Fibonacci design to receive MSI-1436. Drug infusions will last approximately 2 hours. If a subject has a dose-limiting toxicity (DLT) at any time during the study, MSI-1436 will be held and either re-started or discontinued in that subject as per the Dose Adjustments and Toxicities Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Signed, witnessed, and dated Institutional Review Board (IRB) approved Informed Consent Form (ICF).
* Pathologically confirmed metastatic breast cancer with measurable disease. Metastatic sites must be measurable on CT, MRI, or FDG-PET/CT as per the revised RECIST v1.1 criteria or measurable disease on physical examination.

A metastatic site must be biopsy proven

* Life expectancy ≥3 months.
* Patients enrolled must have received 2 or more lines of therapy and all patients with HER2 expressing tumors must have received HER2 targeted therapy.
* Female Age ≥18 years.
* Stable brain metastasis is permitted. This is not considered measurable disease.

Stable brain metastasis is defined as no change on CT scan or MRI for minimum of 2 months AND no change in steroid dose for a minimum of 4 weeks

* A negative serum pregnancy test, if female of reproductive potential. Reproductive potential defined as age < 55 or with no menses for < 1 year
* Screening laboratory values as follows:

Total bilirubin ≤1.5 times upper limit of normal (ULN). Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) and alanine aminotransferase (serum glutamic pyruvate transaminase)≤ 2.5 times ULN.

Serum creatinine ≤2.0 mg/dL or calculated creatinine clearance ≥60 mL/min. Absolute neutrophil count >1,500 cells/mm3. Platelet count ≥100,000 plt/mm3. Hemoglobin ≥ 8 g/dL. Non-diabetic

Exclusion Criteria:

* Pregnant or breast-feeding
* ECOG Performance Status greater than 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04; Primary Completion 2017-07 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Maximally Tolerated Dose (MTD) of MSI-1436 | one year
  Subjects will be enrolled according to a standard Phase I Fibonacci design to receive MSI-1436C. If a subject has a dose-limiting toxicity (DLT) at any time during the study, MSI-1436C will be held and either re-started or discontinued in that subject as per the Dose Adjustments and Toxicities Guidelines.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | one year
  The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to drug after administration of a dose of MSI-1436C.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | one year
  All adverse events and dose-limiting toxicities will be recorded and tabulated. A dose-limiting toxicity (DLT) will be defined as any grade 3 or higher NCI Common Toxicity Criteria adverse event (CTCAE) that is deemed related to the study drug MSI-1436C, any infusion reaction necessitating drug discontinuation, or any other drug related adverse event leading to the study drug discontinuation.
  Descriptive statistics will be used to summarize adverse events and dose-limiting toxicities. The proportion of AEs and DLTs will be calculated along with their corresponding exact 95% confidence intervals.
response rates | one year
  To assess the response rates of MSI-1436C in metastatic breast cancer patients the outcome variable of interest is time-to-progression. Patients who have not progressed (or who have not died) as of their last known follow-up, will be considered 'censored' for the time-to-progression analysis.
  Time-to-progression will be estimated using the Kaplan-Meier Product-Limit Method. Any post- hoc group comparisons will be carried out using the log-rank test. Patients who have not progressed (or who have not died) as of their last known follow-up, will be considered 'censored' for the time-to-progression analysis.
Peak plasma concentration of the drug after administration (cmax) | one year
  The maximum (or peak) serum concentration that MSI-1436C achieves in the plasma after the drug has been administrated and prior to the administration of a second dose.
Time to reach cmax | one year
  The amount of time for MSI-1436C to reach Cmax
Time required for the concentration of MSI-1436C to reach half of its original value, or half life (t1/2) | one year
  The time required for the concentration of MSI-1436C to reach half of its original value.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Budman, MD, Principal Investigator — North Shore LIJ Cancer Institute
Locations (1):
- CFAM / Monter Cancer Center, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No